CLINICAL TRIAL: NCT01534455
Title: A Randomized Phase II Study to Determine the Efficacy and Tolerability of Two Doses of Eribulin Plus Lapatinib in Trastuzumab Pre-treated Patients With HER2-positive Metastatic Breast Cancer (E-VITA)
Brief Title: Efficacy and Tolerability of Eribulin Plus Lapatinib in Patients With Metastatic Breast Cancer (E-VITA)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: very slow patient recruitment and concerns about the actuality of the study design
Sponsor: GBG Forschungs GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBG 64; 2010-023237-37 (EudraCT Number)
Record Dates: First submitted 2012-02-08; First posted 2012-02-16 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Metastatic Breast Cancer
Keywords: German Breast Group; GBG Forschungs GmbH; GBG; GBG 64; E-VITA; Breast Cancer; Metastatic Breast Cancer; Eribulin; Lapatinib; Halaven; Tyverb
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lapatinib + 1,23 mg Eribulin (Experimental)
  Interventions: Drug: Lapatinib + 1,23 mg Eribulin
- Lapatinib + 1,76 mg Eribulin (Experimental)
  Interventions: Drug: Lapatinib + 1,76 mg Eribulin

INTERVENTIONS:
Drug: Lapatinib + 1,23 mg Eribulin — Lapatinib 1000 mg/day + Eribulin 1,23 mg/m2 i.v. on day 1 and 8, q21
  Arms: Lapatinib + 1,23 mg Eribulin
Drug: Lapatinib + 1,76 mg Eribulin — Lapatinib 1000 mg/day + Eribulin 1,23 mg/m2 i.v. on day 1 and 8, q21
  Arms: Lapatinib + 1,76 mg Eribulin

SUMMARY:
* Lapatinib in combination with capecitabine has been approved for the treatment of women with HER-2-positive advanced breast cancer that have progressed after anthracycline-, taxane-, and trastuzumab-containing therapies. The use of this combination is limited by overlapping toxicity such as diarrhea and cutaneous side effects.
* A significant number of patients receive today capecitabine with trastuzumab as first- or second-line treatment. Therefore, other combinations of lapatinib with less toxic cytotoxic agents are needed.
* Eribulin mesylate (E7389) is a synthetic analog of Halichondrin B (HalB), a large polyether macrolide isolated from a marine sponge. Eribulin is a mechanistically unique antagonist of microtubule dynamics among tubulin-targeted agents, leading to inhibition of microtubule growth in the absence of effects on microtubule shortening, and formation of non- productive tubulin aggregates.
* Eribulin mesylate at a dose of 1.4 mg/m² given on day 1, 8 every 3 weeks has shown better overall survival by 2.5 months compared to treatment of physicians choice in patients with locally advanced or metastatic breast cancer who were previously treated for 2-5 lines with anthracyclines, taxanes, and capecitabine (EMBRACE study).
* The most frequently reported eribulin-related AEs were asthenia/fatigue (65%), alopecia (60%), neutropenia (60%), nausea (44%), anemia (28%), pyrexia (23%), leucopenia (22%), anorexia (21%), constipation (19%), vomiting (18%), and peripheral neuropathy (5.5%; only grade 3). Grade 4 neutropenia occurred in 32% of patients, and febrile neutropenia occurred in 5.5% of patients. The frequency of all other grade 3/4 AEs was less than 3%. This toxicity profile does not overlap with that of lapatinib.
* There is uncertainty in how far a once every 3 week schedule of eribulin mesylate at a dose of 2.0 mg/m² would be better tolerated. Several phase II studies are currently conducted in various non-breast cancer indications to compare the d1+8 q d21 with a d1 q d21 schedule.
* The aim of this randomized phase II study is to compare the efficacy and tolerability of two dose-schedules of eribulin plus lapatinib in HER2-positive breast cancer, pre-treated with trastuzumab in the adjuvant and/or metastatic setting.

DETAILED DESCRIPTION:
Primary Objectives

1. To assess the time to progression (TTP) of eribulin at a dose of 1.23 mg/m² IV days 1+8, q 21 and eribulin given at a dose of 1.76 mg/m² IV day 1, q d21 both in combination with lapatinib.
2. To assess the safety and toxicity of both treatment arms.

Secondary Objectives

1. To determine the objective response rate of both treatment arms.
2. To determine the overall clinical benefit rate (CR + PR + SD >24 weeks) of both treatment arms.
3. To determine overall survival in both treatment arms 3 years after 1st patient has been randomized.
4. To assess biomarkers like PI3K mutation, PTEN expression, c-myc on the primary tumor and correlate them with TTP in both treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to beginning specific protocol procedures, including expected cooperation of the patients for the treatment and follow-up, must be obtained and documented according to the local regulatory requirements.
* Complete baseline documentation must be submitted via the web-based data collection system MedCODES® to the GBG Forschungs GmbH.
* Histological confirmed carcinoma of the breast with over-expression of HER2 (IHC3+ or FISH pos., according to current guidelines of AGO). Every effort should be made to make paraffin embedded tissue or slides from the original tumor and/or from metastatic tissue available for confirmation of diagnosis and additional translational research.
* Locally advanced or metastatic stage of disease not suitable for surgery or radiotherapy alone.
* Patients must have either measurable or non-measurable target lesions according to RECIST criteria. Complete staging work-up within 4 weeks prior to registration. All patients must have chest X-ray (PA and lateral), abdominal ultrasound or CT scan or MRI, and bone scan. In case of positive bone scan, bone X-ray is mandatory. Other tests may be performed as clinically indicated.
* The following previous systemic treatments are eligible:

  * Previous treatment with trastuzumab either as (neo)adjuvant treatment for early breast cancer and/or first and/or second line treatment for metastatic breast cancer,
  * adjuvant and up to 2 chemotherapy regimen for metastatic breast cancer,
  * if previous chemotherapy regimen were anthracycline based, the maximum cumulative dose of prior anthracycline therapy must not exceed 360 mg/m² for doxorubicin and 720 mg/m² for epirubicin,
  * adjuvant endocrine therapy,
  * palliative endocrine treatments,
  * treatment with bisphosphonates (adjuvant and/or palliative),
  * at least 4 weeks since radiotherapy, with full recovery. The measurable disease must be completely outside the radiation field or there must be pathologic proof of progressive disease. 7. Age >18 years. 8. ECOG performance status 0-2. 9. Laboratory requirements:
  * Absolute neutrophil count ≥ 1500 cells/ul,
  * hemoglobin ≥ 10.0 g/dL (hemoglobin <10.0 g/dL is acceptable if it is corrected by growth factor or transfusion),
  * platelet count ≥100,000 cells/ul,
  * bilirubin <= 1.5x the upper limit of normal for the institution (ULN),
  * elevation of transaminases and alkaline phosphatase < 2.5x ULN or <5x ULN for patients with liver metastases,
  * creatinine <= 1.5 x ULN or creatinine-clearance > 40 ml/min (according to Cockroft Gault),
  * negative pregnancy test (urine or serum) within 14 days prior to registration for all women of childbearing potential. 10. Normal cardiac ejection function as determined by cardiac ultrasound (LVEF above institutional normal range).

    11. A female either of:
* Non-childbearing potential i.e., physiologically incapable of becoming pregnant because of history of hysterectomy, bilateral oophorectomy (ovarectomy), bilateral tubal ligation or postmenopausal status.
* Childbearing potential with a negative serum pregnancy test within 2 weeks prior to registration, preferably as close to the first dose as possible, and agrees to use adequate contraception. Acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follow:

  * An intrauterine device with a documented failure rate of less than 1% per year.
  * Vasectomized partner who is sterile prior to the female subject's entry and is the sole sexual partner for that female.
  * Complete abstinence from sexual intercourse for 14 days before exposure to investigational product, through the dosing period, and for at least 21 days after the last dose of investigational product.
  * Double-barrier contraception (condom with spermicidal jelly, foam suppository, or film; diaphragm with spermicide; or male condom and diaphragm with spermicide). 12. Female patients who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug.

    13. Patients must be available and compliant for treatment and follow-up. Patients registered on this trial must be treated and followed up at the participating or a cooperating center.

Exclusion Criteria:

* Known hypersensitivity reaction to the compounds or incorporated substances (e.g. halichondrin B and/or halichondrin B chemical derivative).
* Patients who have received eribulin or lapatinib before.
* Concurrent immunotherapy or hormonal therapy (anti-hormonal, contraceptive and/or replacement therapy). Bisphosphonates may be continued.
* Life expectancy of less than 3 months.
* Parenchymal brain metastases, unless adequately treated by neurosurgery, radiotherapy, radiosurgery or a combination.
* Any ongoing toxicity from prior anti-cancer therapy that is grade >1 and/or that is progressing in severity, except alopecia or for stable sensory neuropathy Grade 2.
* Known or suspected congestive heart failure (>NYHA I) and/or coronary heart disease, angina pectoris requiring anti-anginal medication, previous history of myocardial infarction, evidence of transmural infarction on ECG, un- or poorly controlled arterial hypertension (i.e. BP >150/100 mmHg under treatment with two antihypertensive drugs), rhythm abnormalities requiring permanent treatment, clinically significant valvular heart disease.
* Currently active infection.
* History of other malignancies within the last 5 years which could affect the diagnosis, assessment or prognosis of metastatic breast cancer.
* Malabsorption syndrome or insufficient gastrointestinal function, preexisting diagnosis of ulcerative colitis.
* Concurrent treatment with other experimental drugs; participation in another clinical trial with any investigational not marketed drug within 30 days prior to study entry.
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Time to Progression (TTP) | 3 years
Safety of the Therapy | 3 years
  Number and percentage of participants who comply and tolerate the Therapy.
Toxicity of Therapy | 3 years
  Number and percentage of participants with Adverse Events (any Grade and Grade 3/4).

SECONDARY OUTCOMES:
Objective Response Rate | 3 years
Overall Clinical Benefit Rate | 3 Years
Overall Survival | 3 Years
Assess PI3K mutation, PTEN expression and c-myc (Biomarkers) on primary tumor | 3 Years
  Correlate the PI3K mutation, PTEN expression and c-myc found in the FFPE tissue samples with primary tumor characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Bischoff, MD, Principal Investigator — University Women's Hospital Magdeburg
Locations (1):
- Klinikum der Otto-v.-Guericke-Universität Frauenklinik, Magdeburg, Germany